CLINICAL TRIAL: NCT02694068
Title: Biological Determinants of Peritoneal Dialysis
Acronym: Bio-PD
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Rajnish Mehrotra, Dr. Rajnish Mehrotra, MD. Professor of Medicine, Division of Nephrology, University of Washington, University of Washington
Other Study IDs: STUDY00002027
Record Dates: First submitted 2016-02-12; First posted 2016-02-29 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: End-Stage Kidney Disease
Keywords: Peritoneal Dialysis; Genetic; Peritoneal Membrane; Peritoneal Equilibrium Test; Ultrafiltration Capacity; End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, Dialysate, and DNA may be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Discovery for Aim One: 2173 subjects will be involved in the discovery cohort.
  Interventions: Other: Peritoneal Equilibrium Test; Other: 4 hour dwell of 2.5/4.25% dextrose solution
- Replication for Aim One: 1673 subjects will comprise the replication cohort.
  Interventions: Other: Peritoneal Equilibrium Test; Other: 4 hour dwell of 2.5/4.25% dextrose solution
- Discovery for Aim Two: 824 subjects will be involved in the discovery cohort.
  Interventions: Other: Peritoneal Equilibrium Test; Other: 4 hour dwell of 2.5/4.25% dextrose solution
- Replication for Aim Two: 538 subjects will comprise the replication cohort.
  Interventions: Other: Peritoneal Equilibrium Test; Other: 4 hour dwell of 2.5/4.25% dextrose solution

INTERVENTIONS:
Other: Peritoneal Equilibrium Test — These will be done as part of standard of care procedures. PETs will not be performed solely for research purposes.
Other: 4 hour dwell of 2.5/4.25% dextrose solution — If a PET is not performed annually as part of standard of care, subjects will undergo a 4 hour timed dwell with either 2.5 or 4.25% dextrose solution. This will be for the purposes of sample collection and/or measurement of ultrafiltration capacity.

SUMMARY:
Peritoneal Dialysis (PD) is a technique for treating kidney failure where fluid is instilled into the body's peritoneal cavity. Fluid and solutes travel across the peritoneal membrane, and the function of this membrane is critical to successful PD. Studies have shown that certain demographic and clinical variables explain a very small part of the variability in baseline function. This study will further explore the common genetic variants that determine the baseline peritoneal membrane function in patients starting treatment with PD and change in function upon treatment .

This study will incorporate data from subjects' first ever peritoneal equilibrium test (PET), changes in the transfer of water across the peritoneal membrane over time, demographic information, and results from laboratory analysis of DNA, blood, and dialysate. The investigators hope that this study will provide information on the biological pathways that account for variability in the peritoneal membrane. This could ultimately lead to the development of biomarkers to identifying individuals at risk for decline in peritoneal membrane function over time and/or be used to identify novel therapeutic targets to preserve or enhance membrane function. Identifying the biological pathways will also increase the understanding of vascular biology, angiogenesis, and fibrosis that could be applied to other tissues and other diseases.

DETAILED DESCRIPTION:
This study will comprise of patient populations from pre-existing biorepositories and prospectively enrolled subjects. DNA will be analyzed from cohorts with data and DNA already collected and available, while prospective sites will collect plasma, DNA, and spent dialysate for further analysis. Clinical data related to the subjects' first ever Peritoneal Equilibrium Test (PET), demographic information, change in ultrafiltration capacity over time, will be correlated with various genetic markers of interest.

Blood and dialysate will be collected at the first study visit, and there will be no additional sample collection. These samples will be collected as part of a PET during a standard of care study visit, or during a timed 4 hour dwell of 2.5% or 4.25% dextrose solution. Annually, subjects will either undergo a PET as standard of care or perform an additional 4 hour dwell as part of the study. These subsequent measures will be utilized to determine change in ultrafiltration capacity over time.

This study has two specific aims:

Aim 1: To identify and validate genetic loci that influence the peritoneal solute transfer rate (PSTR) at start of PD.

Aim 2: To identify and validate genetic loci in pre-specified biologic pathways with change in peritoneal ultrafiltration capacity.

If subjects grant permission, Genome Wide Association Studies (GWAS) results may be transferred to the NIH database of genotypes and phenotypes (dbGaP). Additionally, subjects may agree that remaining samples will be maintained at the University of Washington Kidney Research Institute in a repository for use in future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 20 who are able to provide consent
* Record of a PET within 6 months of starting PD treatment

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing maintenance Peritoneal Dialysis therapy.
Sampling Method: Non-Probability Sample
Enrollment: 4865 (Estimated)
Dates: Start 2015-09-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Four-hour Dialysate to Plasma ratio of creatinine | Prior to study participation or within 6 months of enrollment
  From Peritoneal Equilibration Test performed at the time of start of PD
Change in peritoneal ultrafiltration capacity over time | Once per year (up to 3 years)
  This will be determined from annual assessments of the peritoneal ultrafiltration capacity with a four-hour timed dwell with 4.25%/2.5% dextrose.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanaway IB, Costa IPD, Davies SJ, Perl J, Lambie M, Morelle J, Jarvik GP, Jain AK, Himmelfarb J, Heimburger O, Johnson DW, Pirkle J, Robinson B, Stenvinkel P, Yee-Moon Wang A, Devuyst O, Mehrotra R; Bio-PD Consortium. Genetic Variation and Ultrafiltration with Peritoneal Dialysis: A Genome-Wide Association Study. J Am Soc Nephrol. 2026 Jan 1;37(1):49-66. doi: 10.1681/ASN.0000000803. Epub 2025 Jul 16. PMID 40669005